CLINICAL TRIAL: NCT06663163
Title: The Association Between Fever and CDKL5 Deficiency Disorder: a Nationwide Survey
Status: Completed | Type: Observational
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Principal Investigator, Liankun_Ren, Professor, Xuanwu Hospital, Beijing
Other Study IDs: 2024-127-002
Record Dates: First submitted 2024-10-27; First posted 2024-10-29 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: CDKL5 Deficiency Disorder
Keywords: CDKL5; Drug Resistant Epilepsy; Survey Research
MeSH Terms: conditions — CDKL5 deficiency disorder; Drug Resistant Epilepsy | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observation — This study was an observational study without intervention

SUMMARY:
The primary objective of this research is to study the effects of fever on seizure activity in patients with CDKL5 deficiency disorder

DETAILED DESCRIPTION:
The survey aimed to gather information on seizure during and after fever and hot temperature bath therapy from families of children diagnosed with CDKL5 deficiency disorder through the WeChat group. It is expected to to develop new intervention strategies to reduce seizure frequency, improve patient quality of life, and ultimately address the therapeutic challenges faced by the global CDKL5 patient community.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of CDKL5 deficiency, including molecular confirmation of a pathogenic or likely pathogenic CDKL5 variant and refractory seizures.
* Parents or guardians are willing to complete and provide information about the child's medical history and fever history after receiving the survey questionnaire online.

Exclusion Criteria:

* Any history of previous brain disease (trauma, etc.) that likely to precipitate seizures.
* Presence of any clinical condition that in the opinion of the principal investigator makes the patient not suitable to participate in the trial.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Male or female children with a diagnosis of CDKL5 deficiency, including molecular confirmation of a pathogenic or likely pathogenic CDKL5 variant and refractory seizures.
Sampling Method: Non-Probability Sample
Enrollment: 131 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-12-15 (Actual); Study Completion 2024-12-15 (Actual)

PRIMARY OUTCOMES:
Seizure frequency | Fever episodes within one year leading up to 2 hours of questionnaire completion
  The results of seizure reduction reported in the questionnaire completed by the parents or the seizure diary provided online

CONTACTS AND LOCATIONS:
Overall Officials: Liankun Ren, MD, Principal Investigator — Xuanwu Hospital, Beijing
Locations (1):
- Xuanwu Hospital,Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No